CLINICAL TRIAL: NCT02809417
Title: Interest of the Use of the Web Platform LICORNE (LIaison and COoRdination With a NumériquE Health Reseau) Concerning Coordination of Care for Dependant Elderly Patients
Acronym: LICORNE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 14-PP-17
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Polypathology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- LICORNE platform
- Control

SUMMARY:
This project is associating partners from the public area (university hospital of Nice, Nice university) and the private area (Agfa Health Care, Radhuis, Domicalis) to create a unique medico-psycho-social shared record.

The purpose of this project is to significantly improve coordination of care, especially between hospital and home. We can expect a significant improvement in the patient's living conditions, improving its management, its security and ultimately, lower health care costs.

DETAILED DESCRIPTION:
The LICORNE project was created to give the possibility for the medical establishments to share there medico-psycho-social informations with all actors taking part of the patient care. Indeed, current informatique systems in medical establishments have an isolated functionning, without transmission of information outsite the wall of the hospital. The idea of this project is to bring together all actors involved in the care of a patient around a single shared patient record, regardless of the structures where professionnals work. This project is associating partners from the public area (university hospital of Nice, Nice university) and the private area (Agfa Health Care, Radhuis, Domicalis) to create a unique medico-psycho-social shared record. The informations will be share between all the professionnal taking car of the patient.

The main objective of this protocol will be to determine the impact of using the LICORNE platform on the coordination of care of elderly patients with multiple diseases. We will assess the impact of using the LICORNE platform on the implementation of electronic health record (Dossier Médical Partagé, public health insurance of the social security), and the benefit of using the LICORNE platform to reduce patient's hospital readmissions.

The purpose of this project is to significantly improve coordination of care, especially between hospital and home. We can expect a significant improvement in the patient's living conditions, improving its management, its security and ultimately, lower health care costs.

ELIGIBILITY:
Inclusion Criteria:

* Age> 60 years
* multiple pathologies : having at least two active chronic conditions.
* Polypharmacy : having at least 4 different molecules in its treatment.
* Dependence : GIR 4 or equivalent and less before hospitalization.
* Need medical care at home at least 5 days a week .
* Patient requiring social intervention ( this criterion of judgment is left to the social worker in the patient's file)

Exclusion Criteria:

* Life threatening pathology during current hospitalization .
* Patients undergoing a hospitalization home service .
* Patients without administrative or judicial freedom if the authorization of the legal representative can not be collected.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: old patient with polypathologies and loss of autonomy
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2016-01-28 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2017-01-05 (Actual)

PRIMARY OUTCOMES:
Improvment of the coordinnation around the patient defined by a change of at least one point on a 6 points Likert scale | 6 months

SECONDARY OUTCOMES:
Increase of the number of DMP for the patient using the plateform. Decrease of early hospital readmission | > 15 days
Increase of the number of DMP for the patient using the plateform. Decrease of late hospital readmission | 1 month
Decrease of the time ration hospital/home during the 6 month experimentation | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France